CLINICAL TRIAL: NCT02955238
Title: San Diego Partnership to Reduce Diabetes & Cardiovascular Disease in Latinos
Brief Title: Latinos Understanding the Need for Adherence
Acronym: LUNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Gregory Talavera, Professor & Division Head-Health Promotion/Behavioral Science Graduate School of Public Health, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G00007349
Record Dates: First submitted 2012-07-17; First posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Atherosclerosis; High Blood Pressure; Type 2 Diabetes Mellitus; Heart Disease; Hypercholesterolemia
Keywords: Intervention; Cardiovascular Disease; CVD; Diabetes; Latinos; CIMT; Medication Adherence; Risk Factors; T2D
MeSH Terms: conditions — Atherosclerosis; Hypertension; Diabetes Mellitus, Type 2; Heart Diseases; Hypercholesterolemia; Cardiovascular Diseases; Diabetes Mellitus; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Special Intervention (Experimental): The Special Intervention (SI) is designed to modify multiple, modifiable CVD risk factors that affect atherosclerosis and can be measured by sonography of the carotid intimal thickness. The SI is designed to address multiple, modifiable CVD risk factors that involve medication therapy, including hypertension, diabetes, and dyslipidemia.
  Interventions: Behavioral: Special Intervention
- Usual Care (No Intervention): Usual care (UC) reflects current practices by the primary care providers in the adult medicine department. Participants randomized into the UC group will continue with their regular medical visits and referrals to the health educator as they were before randomization.

INTERVENTIONS:
Behavioral: Special Intervention — Participants randomized into the SI group will participate in four group health education classes and seven clinical visits per year with the "patient care team". The patient care team will be comprised of a mid-level clinician and a Community Health Worker (CHW).
  Content and materials utilized in the group health education classes are derived from the validated and translated curriculum Pasos Adelante , developed and refined by the CDC. Methods for training CHWs will be derived from the Pasos Adelante Curriculum.
  Arms: Special Intervention

SUMMARY:
The Latino population in the United States is increasing in size; is diverse in culture, backgrounds and countries of origin; is experiencing unique influences from social and behavioral acculturation to the U.S.; is reported nationally to have lower rates of heart disease; is reported to have increased prevalence of diabetes and asthma; and is generally poorer and less educated (NHLBI working Group, 2003). They represent an important target population for disparities research. In particular Latinos accessing care in Community Health Centers in the United States represent an ideal population for conducting disparities research because lack of access to care is minimized through various governmental health insurance support mechanisms. This study will build on existing relationships to conduct the proposed study, using expertise in epidemiologic, behavioral and genetic research in an effort to promote a coordinated, comprehensive, interdisciplinary and focused research effort to improve the care being delivered to indigent Latinos at-risk for and with CVD.

DETAILED DESCRIPTION:
This study will build on existing relationships to conduct the proposed study, using expertise in epidemiologic, behavioral and genetic research in an effort to promote a coordinated, comprehensive, interdisciplinary and focused research effort to improve the care being delivered to indigent Latinos at-risk for and with cardiovascular disease (CVD). This study consists of three study visits:

Study Visit 1 (Sv1):

During Sv1, which lasts about 2 hours, potential participants are recruited and the consenting process is completed with those who wish to take part in the study. Participants then have their blood pressure taken and blood draw takes place. After the blood draw participants will be given a snack before completing the battery of psychosocial, health history and risk factor questionnaires. Lastly, standing height, weight and bioelectric impedance (Tanita scale) will be measured to determine BMI/obesity as a risk factor. At the end of Sv1 participants will be given the GT3X actigraph to objectively monitor their physical activity. Participants will be asked to wear the activity monitor for seven days and asked to return the monitor at the Sv3 appointment.

Chart Audit:

A chart audit will be performed by a research assistant (RA) before Sv3 in order to confirm eligibility and confirm medical history. Information from the chart may also lead to exclude individuals with deteriorated health status. If such a condition is detected the investigators will consult with the primary care provider for confirmation and adjudication before notifying the patient.

Study Visit 2 (Sv2):

The second study visit will take place in the form of a telephone call. After Sv1 a member of the research team will call participants to confirm eligibility and continued interest in the randomized controlled trial. If participants are still interested and eligible, they will continue with Sv3.

Study Visit 3 (Sv3):

The final study visit and randomization will take place at the LUNA field site, where the B-mode ultrasound machine will be stationed. During this time participants will have 1) the Carotid Intimal Medial Thickness (CIMT), the primary outcome, measured using non-invasive ultrasonography, 2) the difference in blood pressure between legs and arms, called Ankle Brachial Index (ABI), and 3) complete any outstanding/incomplete questionnaires from Sv1. During SV-3 the informed consent will be reviewed one more time. The physical measures of CIMT and ABI will be performed by trained technicians.

Also during Sv3, participants will be provided with Medication Event Monitoring System (MEMS) tracking caps. These caps will be used to objectively monitor participant adherence to their recommended chronic disease medications, either their lipid lowering, hypertensive or diabetes medication. In both groups it will provide the study with objective information on medication use behavior and for the intervention group the information serve as feedback to improve adherence to pill taking behavior.

Both control and experimental conditions will be asked to participate in the medication adherence study component, which will begin immediately after study group randomization. Participants' medication adherence will be monitored for one year including four prescription refill time points.

In addition to completing the comprehensive baseline assessments during SV-1 through SV-3, the extended screening period allows the participant time to consider and discuss their participation in the study. If participants have less than one defined CVD risk factors or refuse to participate in the RCT, they will be offered participation in the observational study (i.e. study in which only base-line measures and subsequent routine measures obtained during usual care will be analyzed). The observational group will serve as another comparison group for the overall chronic disease study.

ELIGIBILITY:
Inclusion Criteria:

1. be of Hispanic/Latino ethnicity
2. be a registered patient at the SYHC, Inc.
3. be at least 40 years of age or older
4. have one or more modifiable CVD risk factors, which are defined here as: high LDL cholesterol (non-diabetic threshold = > 160 mg/dl, diabetic threshold = > 130 mg/dl), low HDL cholesterol (<40 mg/dl), Obesity (BMI > 30 kg/m2), Cigarette smoking (daily smoker), Diabetes (fasting blood glucose > 126, self-reported and/or confirmed from chart review), and Hypertension (BP > 140/90 mmHg, or on hypertensive meds); and 5) not be currently participating in any other CVD program.

Exclusion Criteria:

1. are pregnant (temporary exclusion-may qualify six months post partum)
2. planning to move out of the area in the next six months
3. have health problems, disabilities, or mental problems so severe as to prohibit informed consent and actual clinic/special intervention attendance. The most common abnormality that will be found on the ultrasound scans (CIMT) is extensive carotid disease. For some individuals, this may make examination of the carotid arteries very difficult. Thus, individuals will be excluded if 4) there is extensive carotid disease that precludes an accurate assessment of CIMT.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2009-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Carotid Intimal Medial Thickness (CIMT) Measurement | Baseline and 24-months
  The CIMT measurement measures the thickness of the inner two layers of the carotid artery. The special intervention arm of this randomized trial is designed to modify multiple, modifiable cardiovascular risk factors that affect atherosclerosis and can be measured by sonography of the carotid intimal thickness.

SECONDARY OUTCOMES:
Medication Adherence | Baseline and every 6-months for a maximum of 2-years
  Medication adherence in measured using Medication Event Monitoring System (MEMS caps)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Talavera, MD/MPH, Principal Investigator — San Diego State University
Locations (1):
- South Bay Latino Research Center, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No